CLINICAL TRIAL: NCT02262013
Title: Evaluation of a Family-based Pediatric Obesity Program: TEENS+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM20003076
Record Dates: First submitted 2014-10-07; First posted 2014-10-10 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Pediatric Obesity
Keywords: Pediatric Obesity; Lifestyle Intervention; Family-based Intervention; Motivational Interviewing
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parents as Coaches (Active Comparator): PAC (modeled after NIH-funded NOURISH) focuses on parenting strategies to support and facilitate their child's weight management via family-based change. Each visit includes group psychoeducation and discussion, focused on parenting strategies to facilitate healthy weight management in their child(ren). Topics include focus such as role modeling, strategies for healthy lifestyle changes, and how to be a coach to your teen.
  Interventions: Behavioral: Parents as Coaches
- Parent Weight Loss (Experimental): In PWL parents will be given a weight loss goal of 1-2 lbs/week, as well as specific calorie and fat prescriptions, PA goals, and instructions to self-monitor key information. Parents will receive training in core behavioral weight loss strategies (e.g., goal setting, stimulus control) and techniques to help them achieve these goals and will also receive personalized feedback throughout the program.
  Interventions: Behavioral: Parent Weight Loss

INTERVENTIONS:
Behavioral: Parents as Coaches — Adolescents will receive lifestyle intervention (TEENS) and parents will receive parents as coaches (PAC) intervention.
  Other Names: TEENS+PAC
  Arms: Parents as Coaches
Behavioral: Parent Weight Loss — Adolescents will receive lifestyle intervention (TEENS) and parents will receive parent weight loss (PWL) intervention.
  Other Names: TEENS+PWL
  Arms: Parent Weight Loss

SUMMARY:
Investigators propose to pilot an adolescent obesity intervention, TEENS+, to examine the feasibility of this dietary intervention strategy and preliminary effectiveness of two models of parental involvement within adolescent obesity treatment.

DETAILED DESCRIPTION:
Investigators will recruit overweight or obese adolescents (BMI >85th percentile) and parent(s) (BMI >25 kg/m2). Families will participate in one of two 6-month treatments: 1) TEENS+Parents as Coaches (PAC), engaging parents as helpers in their child's weight management, or 2) TEENS+Parent Weight Loss (PWL), engaging parents in their own weight management. All adolescents will participate in TEENS+, which includes behavioral support, nutrition education, and supervised physical activity.

For the adolescents, intervention will consist of weekly 1 hour exercise sessions and alternating weekly 1 hour behavioral and nutrition group sessions. Parents will also attend the nutrition sessions and participate in a behavioral parent-only biweekly group. Parent behavioral group sessions will be specific to the treatment arm (e.g. PAC or PWL). Assessments will consist of anthropometric measures, lab work, psychological surveys, and nutritional evaluations. Assessments will be completed at baseline, 3 months, 6 months (post-intervention), and 9 months.

ELIGIBILITY:
Inclusion Criteria: Overweight (BMI ≥85% percentile for age and gender according to the CDC Growth Charts) males and females between the age of 12 and 17 years will be eligible for study participation. In order to be eligible, the adolescent must also reside with the primary participating parent, who has a BMI ≥25 kg/m 2 and is also willing to participate in the study protocol. Eligible families must live within a 30 mile radius of the Healthy Lifestyles Center (HLC) at Children's Hospital of Richmond (CHoR) at VCU where the interventions will be conducted.

Exclusion Criteria:

Adolescents and parents will be ineligible for study participation under the following conditions: 1) non-English speaking; 2) medical condition(s) that may be associated with unintentional weight change (e.g., hypothalamic injury, Prader-Willi, or malignancy); 3) diabetes mellitus diagnosed by history or a fasting glucose ≥126 mg/dl (subjects with glucose intolerance or "pre-diabetes" will eligible for study participation); 4) use of oral glucocorticoids, atypical antipsychotics, weight loss medications, or an investigational medication within 3 months of study participation; 5) medical condition(s) that may be negatively impacted by exercise; 6) physical limitation affected the ability to exercise, 7) psychiatric, cognitive or developmental conditions that would impair the adolescent's ability to complete assessments or participate in a group; 8) reports of compensatory behaviors (i.e., vomiting, laxative abuse, excessive exercise) in the past 3 months; 9) current pregnancy or plan to become pregnant during study period; 10) previous participation in TEENS or NOURISH; 11) current participation in another weight loss program; or 12) personal history of weight loss surgery.

Adolescents and parents taking metformin, oral contraceptives, tricyclic antidepressants (TCAs), selective serotonin reuptake inhibitors (SSRIs), or stimulant medications may be eligible for participation; however, subjects must be on a stable dose of medication for at least 3 months prior to study participation.

In addition, adolescents will be excluded from participation (and referred for further evaluation) based on the results of baseline psychological assessments under the following circumstances: 1) clinically significant depression, evidenced by elevations (>20) on CDI; 2) suicidality as reported on CDI or during screening / behavioral interview; 3) psychosis, 4) clinical impairment in Activities of Daily Living and Functional Communication (i.e., expressive and receptive communication; and 3) clinically significant eating disorder based on EDE-Q.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2015-01; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in BMI z-scores (adolescents and parents) | 3 months, 6 months, 9 months

SECONDARY OUTCOMES:
Changes in Insulin Sensitivity | 6 months, 9 months
  Insulin, Glucose, HbA1c
Changes in Serum Lipids | 6 months, 9 months
Changes in Energy Balance | 6 months, 9 months
  Adipokines, Cytokines
Changes in Blood Pressure | 3 months, 6 months, 9 months
Changes in Psychosocial Measures | 3 months, 6 months, 9 months
Changes in Dietary Intake | 3 months, 6 months, 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Edmond P Wickham, MD, MPH, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond at VCU Healthy Lifestyles Center, Henrico, Virginia, United States